CLINICAL TRIAL: NCT00436644
Title: A Phase II Trial of Lapatinib in Combination With Weekly Topotecan in Patients With Platinum-Refractory/Resistant Ovarian and Primary Peritoneal Carcinoma
Brief Title: Lapatinib and Topotecan in Treating Patients With Ovarian Epithelial Cancer or Primary Peritoneal Cancer That Did Not Respond to Cisplatin or Carboplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Paul Haluska, M.D., Ph.D., Mayo Clinic Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC0661; P30CA015083 (NIH); RC0661 (Other: Mayo Clinic Cancer Center & MCCRC); 06-002426 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2012-03-22 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Lapatinib; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib + Topotecan (Experimental): Assess biological effects of topotecan and lapatinib in patients with epithelial ovarian cancer and primary peritoneal carcinoma.
  Interventions: Drug: Lapatinib; Drug: Topotecan

INTERVENTIONS:
Drug: Lapatinib — 1250 mg orally days 1 -28.
  Other Names: Tykerb
Drug: Topotecan — 3.2 mg/m2 IV over 30 min in 100mL D5W (5% dextrose in water) or 0.9% NS at days 1, 8 & 15.
  Other Names: Hycamptin

SUMMARY:
RATIONALE: Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving lapatinib together with topotecan may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving lapatinib together with topotecan works in treating patients with ovarian epithelial cancer or primary peritoneal cancer that did not respond to cisplatin or carboplatin.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of lapatinib ditosylate and topotecan hydrochloride, in terms of response, in patients with platinum-resistant or refractory ovarian epithelial or primary peritoneal cavity carcinoma.

Secondary

* Determine the overall survival time in patients treated with this regimen.
* Determine the time to progression in patients treated with this regimen.
* Assess the toxicity profile of this regimen in these patients.

Translational

* Determine the expression patterns of epidermal growth factor receptor, HER2/neu, hypoxia-induced factor 1 alpha, CD31, breast cancer resistance protein, and topoisomerase I by immunohistochemistry using tumor tissue from primary debulking surgery.
* Determine the feasibility of monitoring circulating tumor cells with specific biological markers to determine or follow response in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral lapatinib ditosylate once daily on days 1-28 and topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and on day 8 of course 1 (immediately after the topotecan infusion) and are evaluated for pharmacological studies. Tumor tissue samples obtained at debulking surgery are examined by immunohistochemistry for epidermal growth factor receptor, HER1, ErbB1, HER2/neu, ErbB2, hypoxia-induced factor 1 alpha, CD31, platelet endothelial cell adhesion molecule 1, topoisomerase I, and breast cancer resistance protein.

After the completion of study treatment, patients are followed periodically for 2 years.

PROJECTED ACCRUAL: A total of 39 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial or primary peritoneal carcinoma
* Must have one of the following:

  * Measurable disease
  * Evaluable disease AND a CA-125 value that has increased ≥ 2 times the nadir value established after debulking surgery and first-line chemotherapy, confirmed by a second measurement within the past 21 days

    * If a second measurement has not been done, it can be done ≥ 7 days but < 21 days prior to study treatment
* Platinum-refractory and/or -resistant disease after first-line chemotherapy

  * Patients retreated with platinum agents (i.e., second relapse) are not eligible
  * Patients treated with first-line triplet therapy (e.g., on clinical trial GOG-182) are eligible
* Must have had debulking surgery

  * Tissue blocks from this surgery must be available
* No CNS metastases

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 3 times ULN (5 times ULN if there is liver involvement)
* Creatinine ≤ 1.5 times ULN
* Hemoglobin ≥ 9.0 g/dL
* No uncontrolled infection
* No New York Heart Association class III or IV heart failure
* Left Ventricular Ejection Fraction (LVEF) ≥ 50% by echocardiogram
* No seizure disorder
* No other prior or concurrent malignancy in the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior topotecan hydrochloride
* More than 4 weeks since prior surgery or procedure involving the peritoneum or pleura

  * CA125 measurements used as basis for enrollment must be made outside of this 4-week window
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* More than 4 weeks since prior immunotherapy
* More than 4 weeks since prior biologic therapy
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to > 25 % of bone marrow
* No prior therapy with an anti-epidermal growth factor receptor or anti-HER2 tyrosine kinase inhibitors
* No prior agents targeting topoisomerase I
* No prior or concurrent human anti-mouse antibodies (HAMA) in patients with non-measurable disease
* At least 14 days since prior and no concurrent herbal or dietary supplements

  * Vitamin supplements are allowed unless they include herbal additives
* At least 14 days since prior and no concurrent CYP3A4 inducers, including any of the following:

  * Rifampin
  * Rifabutin
  * Rifapentine
  * Phenytoin
  * Carbamazepine
  * Phenobarbital
  * Efavirenz
  * Nevirapine
  * Cortisone (> 50 mg)
  * Hydrocortisone (> 40 mg)
  * Prednisone (> 10 mg)
  * Methylprednisolone (> 8 mg)
  * Dexamethasone (> 1.5 mg)

    * Oral doses of ≤ 1.6 mg of dexamethasone allowed
  * Modafinil
  * Hypericum perforatum (St. John's wort)
* At least 7 days since prior and no concurrent CYP3A4 inhibitors, including any of the following:

  * Clarithromycin
  * Erythromycin
  * Troleandomycin
  * Itraconazole
  * Ketoconazole
  * Fluconazole (> 150 mg daily)
  * Voriconazole
  * Delaviridine
  * Nelfinavir
  * Amprenavir
  * Ritonavir
  * Indinavir
  * Saquinavir
  * Lopinavir
  * Verapamil
  * Diltiazem
  * Nefazodone
  * Fluvoxamine
  * Cimetidine
  * Aprepitant
  * Grapefruit or grapefruit juice
* At least 6 months since prior and no concurrent amiodarone
* No concurrent participation in another study involving a pharmacologic agent (e.g., drugs, biologics, immunotherapy, gene therapy) for symptom control or therapeutic intent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Haluska, MD, PhD, Study Chair — Mayo Clinic; John K. Camoriano, M.D., Principal Investigator — Mayo Clinic; Candido E. Rivera, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Mayo Clinic in Jacksonville, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighteen patients were enrolled in stage 1 from February 2, 2007 to May 9, 2008.
Period: Overall Study
Arm/Group | Lapatinib + Topotecan
Started | 18
Completed | 15
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib + Topotecan
Number analyzed (Participants) | 18
Age, Customized [Median (Full Range); unit: Years] | 66 [27 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
Primary Tumor Site [Number; unit: participants]
  Ovarian | 16
  Peritoneal | 2
Primary Tumor Status [Number; unit: participants]
  Platinum Resistant | 5
  Platinum Refractory | 13

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete Response (CR) or Partial Response (PR))
Description: Measurable disease patients: measureable disease is defined as at least one lesion whose longest diameter >= 2cm with conventional techniques or >=1cm with spiral CT
  * Confirmed tumor response (complete and partial) as measured by RECIST(Response Evaluation Criteria In Solid Tumors) criteria on 2 consecutive evaluations at least 4 weeks apart.
  * Confirmed tumor response is at least a 30% decrease in the sum of the longest diameter of target lesions and no new lesions.
  Non-measurable disease patients:
  * Decrement in CA125 by > 50%
  * Improvement in other evaluable disease
Time Frame: Two consecutive evaluations at least 4 weeks apart
Measure: Number; unit: participants
Arm/Group | Lapatinib + Topotecan
Number analyzed (Participants) | 18
participants | 1

2. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the number of months from registration to the date of disease progression, with patients who are progression free being censored on the date of their last evaluation.
Time Frame: Time from registration to progression (up to 2 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib + Topotecan
Number analyzed (Participants) | 18
months | 3.5 [1.9 to 3.9]

3. Secondary Outcome: Adverse Event Profile
Description: Number of patients that experienced adverse events (grade 3 or more) as measured by NCI CTCAE (Common Terminology Criteria for Adverse Events) v3.0
Time Frame: Every 4 weeks
Measure: Number; unit: participants
Arm/Group | Lapatinib + Topotecan
Number analyzed (Participants) | 18
participants
  Neutropenia | 7
  Thrombocytopenia | 5
  Anemia | 1
  Leukopenia | 2
  Diarrhea | 4
  Nausea | 1
  Vomiting | 1
  Dehydration | 2
  Hyponatremia | 1
  Rash | 1
  Fatigue | 1

4. Secondary Outcome: Overall Survival
Description: Overall survival time was defined as the number of months from registration to the date of death or last follow-up
Time Frame: Time from Registration to Death or last follow-up (up to 3 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib + Topotecan
Number analyzed (Participants) | 18
months | 15.5 [12.2 to 24.3]

ADVERSE EVENTS:
Arm/Group | Lapatinib + Topotecan
Serious Adverse Events (participants affected / at risk) | 4/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib + Topotecan (N=18)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib + Topotecan (N=18)
Anemia (Blood and lymphatic system disorders) | 7 (13)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (14)
Nausea (Gastrointestinal disorders) | 5 (9)
Vomiting (Gastrointestinal disorders) | 1 (3)
Disease Progression (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (4)
Leukopenia (Investigations) | 5 (7)
Neutrophil count decreased (Investigations) | 16 (43)
Platelet count decreased (Investigations) | 13 (33)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Pain-Bladder (Renal and urinary disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes